CLINICAL TRIAL: NCT07358299
Title: A Comparison of Haemodynamic Effects, as Assessed by Cardiac Output Monitoring, and Complications of Continuous Versus Single-Shot Spinal Anaesthesia for Hip-Fracture Surgery in Patients Over 50 Years of Age
Brief Title: Haemodynamic Effects and Complications of Continuous Versus Single-shot Spinal Anaesthesia for HIP Fracture Surgery
Acronym: CHIPS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre of Postgraduate Medical Education (Other)
Collaborators: Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Rafał Kamiński, MD, PhD, Associate Professor, Chief of the Department of Orthopaedic and Trauma Surgery (Div. Knee Surg & Arthroscopy, Div. General Orthop Trauma, Div. Upper Limb Surg.) at Gruca Orthopaedic And Trauma Teaching Hospital, Centre of Postgraduate Medical Education
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No. 65/2025 of 16 July 2025
Record Dates: First submitted 2025-09-10; First posted 2026-01-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia, Spinal; Hip Fractures
Keywords: Continuous spinal anaesthesia; Late side effects of spinal anaesthesia; Haemodynamic stability; Follow-up care after proximal femoral fractures; Quality of life after proximal femoral fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single-shot spinal anaesthesia (Experimental): Bolus dose of Bupivacaine Spinal 0,5% Heavy
  Interventions: Drug: Bupivacaine Spinal 0,5% Heavy - bolus
- Continuous spinal anaesthesia (Experimental): Dose titration of Bupivacaine Spinal 0,5% Heavy
  Interventions: Drug: Bupivacaine Spinal 0,5% Heavy - titration

INTERVENTIONS:
Drug: Bupivacaine Spinal 0,5% Heavy - bolus — Group 1 (Control Group) will receive single-shot spinal anesthesia with a bolus of 0.5% hyperbaric bupivacaine, with the dose adjusted according to the patient's weight and height to achieve a sensory block up to the T12 dermatome. The operating table will be kept in a neutral position.
  Other Names: Single bolus
  Arms: Single-shot spinal anaesthesia
Drug: Bupivacaine Spinal 0,5% Heavy - titration — Group 2 (Interventional Group) will receive continuous spinal anesthesia administered via a dedicated intrathecal catheter. An initial induction dose of 1 ml of 0.5% hyperbaric bupivacaine will be administered, followed by titrated boluses of 0.5 ml every 15 minutes until a sensory block to the T12 dermatome is achieved. Once the desired block height is established, the anesthetic level will be maintained by administering titrated doses of 0.5-1 ml approximately every hour. The operating table will be kept in a neutral position.
  Other Names: Rose titration
  Arms: Continuous spinal anaesthesia

SUMMARY:
This research project aims to identify a safer method of spinal anaesthesia for elderly patients undergoing surgical stabilisation of proximal femoral fractures.

The study's primary objective is to compare two spinal anaesthesia techniques: the continuous method (investigational), which allows titration of local anaesthetic doses through a catheter placed in the subarachnoid space, and the conventional single-shot bolus injection.

The main hypothesis is that the continuous catheter technique reduces the incidence of intraoperative hypotension and related complications, such as delirium, acute kidney injury, and cardiovascular events.

Beyond haemodynamic stability-assessed through advanced continuous monitoring of cardiac output and vascular resistance-the study will evaluate early and late complications, as well as quality of life up to 24 months post-surgery.

The project is a prospective, randomised, multicentre clinical trial including at least 216 patients over 50 years of age, randomly assigned to one of the two groups.

Proximal femoral fractures are a major and growing global health issue, particularly among geriatric patients with multiple comorbidities. The conventional single-shot spinal anaesthesia, though widely used, carries a high risk of hypotension, potentially leading to delirium, acute kidney injury, stroke, and cardiac events. These complications worsen prognosis, decrease quality of life, and increase mortality.

Most existing studies are over two decades old, based on small cohorts and outdated anaesthetic protocols, and lack long-term follow-up data (>30 days) on neurological outcomes, functional recovery, quality of life, and mortality. Moreover, no modern trials have provided direct, comprehensive comparisons between single-shot and continuous spinal anaesthesia.

This project therefore seeks to fill this critical evidence gap through a robust randomised clinical trial. Using precise, continuous measurements of arterial pressure, vascular resistance, and cardiac output, alongside long-term assessments of neurological outcomes, quality of life, and survival, it aims to determine whether continuous spinal anaesthesia offers superior safety and should become the new standard of care for this vulnerable population.

DETAILED DESCRIPTION:
Study Flow Diagram.

1. Measured Variables, Measurement Scales, and Tools:

   * Orthopedic and Anesthesiological Qualification: Conducted according to the standard of care and existing procedures at the participating hospital.
   * Baseline Assessment: Performed using the following scales: ASA, Apfel, GCS, RASS, NRS, Bromage, Aldrete, CAM-ICU, and SF-36.
   * Baseline Neurological Assessment: Covering all neurological endpoints specified in the point 7
   * Anesthesia Method (determined by group randomization):

     1. Both groups: Ultrasound-guided femoral nerve block with 10 ml of 0.5% ropivacaine.
     2. Group 1 (Interventional): Continuous spinal anesthesia with titrated doses of 0.5% hyperbaric bupivacaine via an intrathecal catheter. An initial 1 ml induction dose will be administered, followed by 0.5 ml boluses every 15 minutes to achieve a sensory block to the T12 level. Once the block is established, the anesthetic level will be maintained with titrated doses of 0.5-1 ml approximately every hour. The operating table will be kept in a neutral position.
     3. Group 2 (Control): Single-shot spinal anesthesia with a bolus of 0.5% hyperbaric bupivacaine, with the dose adjusted according to the patient's weight and height to achieve a sensory block to the T12 level. The operating table will be kept in a neutral position.
2. Intraoperative Monitoring of Vital Signs:

   1. Standard Monitoring: Continuous measurement of heart rate (HR) via ECG and arterial oxygen saturation (SpO2) via pulse oximetry, as well as non-invasive blood pressure (NIBP) measured at 3, 5, and 15-minute intervals.
   2. Advanced Monitoring: Continuous invasive blood pressure (IBP); uncalibrated cardiac output (CO) measurement-calibrated with stroke volume (SV) calculated by echocardiography (LVOT x VTI*); and continuous measurement of stroke volume variation (SVV), pulse pressure variation (PPV), and systemic vascular resistance (SVR) throughout the intraoperative period.

      * Calculated as the product of the left ventricular outflow tract (LVOT) area and the velocity time integral (VTI), measured in the parasternal long-axis and apical 5-chamber views, respectively.
3. Monitoring in the Post-Anesthesia Care Unit (PACU):

   1. Continuation of standard vital signs monitoring (HR, BP, SpO2).
   2. Continuation of advanced hemodynamic monitoring if hemodynamic instability requires a continuous vasopressor infusion; patients will be transferred to the ICU if stabilization is not achieved.
   3. At discharge from PACU: Assessment using the GCS, RASS, NRS, Aldrete, CAM-ICU, and SF-36 scales, and a neurological assessment covering all endpoints specified in in the point 7 .
4. Monitoring on the Orthopedic Ward:

   a. At hospital discharge: An SF-36 assessment and a neurological assessment covering all endpoints specified in in the point 7 .
5. Assessment of Other Complications: The incidence of other in-hospital complications will be assessed according to established diagnostic criteria if they are suspected to have occurred.
6. Follow-up: Conducted at 1, 3, 6, 12, and 24 months post-intervention. A telephone interview will be performed to complete the SF-36 scale and conduct a neurological assessment covering all endpoints specified in the point 7 .
7. Complications associated with spinal anesthesia:

   1. Postoperative nausea and vomiting (PONV)
   2. Hypothermia
   3. Total spinal anesthesia
   4. Cardiac arrest
   5. Bladder dysfunction
   6. Back pain
   7. Transient neurological symptoms (TNS)
   8. Post-dural puncture headache (PDPH)
   9. Headache other than PDPH
   10. Peripheral nerve palsy
   11. Cauda equina syndrome
   12. Spinal hematoma or hygroma
   13. Intracranial hypotension syndrome
   14. Central nervous system infection
   15. Other

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years, regardless of gender
* Diagnosis of a proximal femur fracture
* Orthopedic qualification for open reduction and internal fixation of the fracture
* Informed consent for the surgical procedure
* Informed consent for regional anesthesia, i.e., a central neuraxial block (spinal anesthesia)
* Informed consent to participate in the study

Exclusion Criteria:

* Age < 50 years, regardless of gender
* Refusal to consent to surgical treatment
* Refusal to consent to regional anesthesia
* Refusal to consent to participate in the study
* Inability to provide informed consent
* Allergy to local anesthetic agents
* Severe congenital or acquired coagulation disorders
* Failure to meet the recommended time interval between the last dose of an anticoagulant and central neuraxial blockade, according to the 2022 European Journal of Anaesthesiology (EJA) guidelines
* Infection at the block site or a systemic infection (i.e., sepsis, septic shock)
* Patients with multiple organ dysfunction syndrome requiring hospitalization in the Intensive Care Unit for stabilization of vital functions
* Clinical signs of increased intracranial pressure or suspicion of an intracranial mass on imaging studies
* Other contraindications to spinal anesthesia as judged by the qualifying physician

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Mild hypotension | periprocedural
  A comparison of frequency and duration of mild hypotensive episodes, defined as a 20% decrease in systolic arterial pressure (SAP) from the baseline value, between spinal anesthesia administered via catheter-based titration dosing (the investigational method) and single-shot administration (the conventional method)

SECONDARY OUTCOMES:
Severe hypotension | periprocedural
  A comparison of frequency and duration of severe hypotension episodes, defined as a decrease in systolic arterial pressure (SAP) of 30% from the baseline value
Hypotension associated with organ complications | periprocedural
  Comparison of the incidence and duration of hypotensive episodes associated with organ complications, defined as a 50% decrease in mean arterial pressure (MAP) from the baseline value
Advanced hemodynamic measurements | periprocedural
  A comparison of the incidence and duration of decrease or increase in the following hemodynamic parameters from their baseline values: cardiac index, CI [ l/min/m²] , stroke volume index, SVI [ml/m²], stroke volume variation index, SVV [%] , pulse pressure variation, PPV [ %], and systemic vascular resistance index, SVRI [ dyn·s·cm-⁵/m²].
  The hemodynamic parameters will be indexed for body surface area
Bradycardia | periprocedural
  Comparison of the incidence and duration of relative and absolute bradycardia, defined respectively as a heart rate (HR) below 60 and 40 beats per minute
Hypotension-related complications | through hospitalisation completion, an average of 1 week
  Comparison of the risk of hypotension-related complications between the study groups:
  1. Delirium
  2. Acute kidney injury (AKI)
Length of stay | through hospitalisation completion, an average of 1 week
  Comparison of the length of stay in the Post-Anesthesia Care Unit (PACU) and Intensive Care Unit (ICU), as well as the total hospital length of stay, between the study groups
Mortality | 0, 1mth, 3mth, 6mth, 12mth, 24mth
  Comparison of the risk of mortality at 1, 3, 6, 12, and 24 months between the study groups
Complications associated with spinal anesthesia: | From admission to the hospital to the end of the 2-year follow-up period
  Comparison of the risk of complications associated with spinal anesthesia:
  1. Postoperative nausea and vomiting (PONV)
  2. Decrease in body temperature / Hypothermia
  3. Total spinal anesthesia
  4. Cardiac arrest
  5. Bladder dysfunction
  6. Back pain
  7. Transient neurological symptoms (TNS)
  8. Post-dural puncture headache (PDPH)
  9. Headache other than PDPH
  10. Peripheral nerve dysfunction
  11. Cauda equina syndrome
  12. Spinal hematoma or hygroma
  13. Intracranial hypotension syndrome
  14. Central nervous system infection
  15. Other
Cardiovascular events | through hospitalisation completion, an average of 1 week
  A comparison of the risk of cardiovascular events (ischemic stroke, acute coronary syndrome) during hospitalization between the study groups
Other complications associated with the studied types of anesthesia | 0 month, 1 month, 3 month, 6 month, 12 month, 24 month
  Comparison of the risk of other complications associated with the studied types of anesthesia
Bromage motor blockade score | periprocedural
  Comparison of the efficacy of both anesthetic techniques, as measured by the degree of motor blockade using the Bromage scale.
  Intensity of motor block, Modified Bromage score (Breen TW 1993)
  1. Complete block (unable to move feet or knees)
  2. Almost complete block (able to move feet only)
  3. Partial block (just able to move knees)
  4. Detectable weakness of hip flexion while supine (full flexion of knees)
  5. No detectable weakness of hip flexion while supine
  6. Able to perform partial knee bend
Minimal clinically important difference | 0 month, 1 month, 3 month, 6 month, 12 month, 24 month
  Assessment of the minimal clinically important difference (MCID) for patient-reported outcome measures (PROMs) to determine the value and extent of clinical improvement and the associated level of patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Rafał Kamiński, MD, PhD, Study Chair — Dept of Musculoskeletal Trauma Surg and Orthop, Gruca Orthopaedic and Trauma Teaching Hospital, CMKP; Magdalena Fleming, MD, Principal Investigator — Dept of Anesthesiology, Gruca Orthopaedic and Trauma Teaching Hospital, CMKP
Locations (2):
- Poland (2):
  - Centre of Postgraduate Medical Education, Professor A. Gruca Teaching Hospital, Konarskiego 13 street, Otwock
  - National Medical Institute of the Ministry of the Interior and Administration, Wołoska 137 street, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raichandani K, Agarwal S, Jain H, Bharwani N. Mortality profile after 2 years of hip fractures in elderly patients treated with early surgery. J Clin Orthop Trauma. 2021 Apr 15;18:1-5. doi: 10.1016/j.jcot.2021.04.009. eCollection 2021 Jul. PMID 33936949
- [Background] Favarel-Garrigues JF, Sztark F, Petitjean ME, Thicoipe M, Lassie P, Dabadie P. Hemodynamic effects of spinal anesthesia in the elderly: single dose versus titration through a catheter. Anesth Analg. 1996 Feb;82(2):312-6. doi: 10.1097/00000539-199602000-00017. PMID 8561333
- [Background] Minville V, Fourcade O, Grousset D, Chassery C, Nguyen L, Asehnoune K, Colombani A, Goulmamine L, Samii K. Spinal anesthesia using single injection small-dose bupivacaine versus continuous catheter injection techniques for surgical repair of hip fracture in elderly patients. Anesth Analg. 2006 May;102(5):1559-63. doi: 10.1213/01.ane.0000218421.18723.cf. PMID 16632842
- [Background] Koole C, Bleeser T, Hoogma DF, Coppens S, Teunkens A, Rex S. Haemodynamic effects of continuous spinal anaesthesia versus single-shot spinal anaesthesia or general anaesthesia for hip fracture surgery: a systematic review and meta-analysis. Br J Anaesth. 2024 May;132(5):1160-1162. doi: 10.1016/j.bja.2023.12.012. Epub 2024 Jan 18. No abstract available. PMID 38242801
- [Background] Viderman D, Aubakirova M, Nabidollayeva F, Abdildin YG. The Analysis of Multiple Outcomes between General and Regional Anesthesia in Hip Fracture Surgery: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Clin Med. 2023 Dec 5;12(24):7513. doi: 10.3390/jcm12247513. PMID 38137582
- [Background] Uppalapati T, Thornton I. Anesthesia Management of Hip Fracture Surgery in Geriatric Patients: A Review. Cureus. 2024 Sep 25;16(9):e70188. doi: 10.7759/cureus.70188. eCollection 2024 Sep. PMID 39463540
- [Background] Barbosa TA, Souza AMF, Leme FCO, Grassi LDV, Cintra FB, Lima RME, Gumieiro DN, Lima LHNE. [Perioperative complications and mortality in elderly patients following surgery for femoral fracture: prospective observational study]. Braz J Anesthesiol. 2019 Nov-Dec;69(6):569-579. doi: 10.1016/j.bjan.2019.09.004. Epub 2019 Nov 11. PMID 31722793
- [Background] Stachurski J, Sionek A. Epidemiology of femoral shaft fractures in Poland. Przegl Epidemiol. 2020;74(3):492-502. doi: 10.32394/pe.74.43. PMID 33576588
- [Background] Wilk R, Skrzypek M, Kowalska M, Kusz D, Wielgorecki A, Horyniecki M, Sliwiak J, Piejczyk S, Pluskiewicz W. Standardized incidence and trend of osteoporotic hip fracture in Polish women and men: a nine year observation. Maturitas. 2014 Jan;77(1):59-63. doi: 10.1016/j.maturitas.2013.09.004. Epub 2013 Sep 14. PMID 24090926
- [Background] Czerwinski E, Kanis JA, Trybulec B, Johansson H, Borowy P, Osieleniec J. The incidence and risk of hip fracture in Poland. Osteoporos Int. 2009 Aug;20(8):1363-7. doi: 10.1007/s00198-008-0787-8. Epub 2008 Nov 14. PMID 19009330
- [Background] Lotan R, Moayad C, Sakhnini M, Rijini N, Goldstein AL, Hershkovich O. In-Hospital Proximal Femoral Fracture Mortality and Anesthesia: Do the First Postoperative 72 h Matter? J Clin Med. 2025 Mar 11;14(6):1885. doi: 10.3390/jcm14061885. PMID 40142693
- [Background] Chatzopoulos ST, Zafeiris CP. Epidemiology of hip fractures in Europe: Geographic variability. Journal of Research & Practice on the Musculoskeletal System (JRPMS). 2023 Dec 1;7(4).